CLINICAL TRIAL: NCT05944328
Title: Effectiveness of a Structured Pharmaceutical Review Intervention of Pharmacotherapeutic Plans to Reduce Medication-related Problems in Geriatric Residences: a Quasi-experimental Pragmatic Assay
Brief Title: Effectiveness of an Intervention of Pharmacotherapeutic Plans to Reduce Medication-related Problems in Geriatric Residences
Acronym: RG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22/191-P
Record Dates: First submitted 2023-06-20; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-03

CONDITIONS: Polypharmacy
Keywords: pharmaceutical intervention; polypharmacy; nursing home

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: systematic and structured review of patient pharmacotherapeutic treatment plans
- control group (No Intervention)

INTERVENTIONS:
Other: systematic and structured review of patient pharmacotherapeutic treatment plans — The intervention consisted of a systematic and structured review of patient pharmacotherapeutic treatment plans to identify problems or situations of risk related to pharmacological treatments and to propose changes or improvements to optimise them. phases:
  Individualised review of pharmacological treatment plans to detect drug-related problems:
  Indication, Appropriateness, Effectiveness, Safety When a drug-related problem was detected according to the above criteria, the pharmacist proposed an adjustment to the pharmacotherapeutic plan. The proposals could include: discontinuation of the drug, change of drug, change to a therapeutic equivalent, initiation of treatment, change of dosage, change of frequency or intensified monitoring.
  The proposals made by the pharmacist were assessed and agreed upon by a committee comprising the doctors responsible and the pharmacist. Thereafter, the consensual proposals for change were discussed with the patient.
  Arms: intervention group

SUMMARY:
Background: Patients living in Geriatric Residences (RG) have increased aging, comorbidity, spending on health resources and mortality. High drug use is associated with an increased risk of falls, disability, and death. It is estimated that 20-50% of inappropriate medications are consumed in the elderly.

Hypothesis: A pharmaceutical intervention based on a clinical review of the pharmacotherapeutic plan of patients in RG will be useful in optimizing the prescription in terms of safety, reducing by 10% or more the inappropriate prescriptions.

Objectives: Evaluate the effectiveness of a structured pharmaceutical intervention based on the clinical review of the pharmacotherapeutic plan to improve its adequacy.

Decrease inadequate prescriptions in patients admitted to RG by 10%

Methodology: Pre-post, quasi-experimental intervention study with control group with prospective follow-up of a cohort of patients in RG. The intervention consists of the clinical review of the pharmacotherapeutic plan carried out by the pharmacist and subsequently agreed in the Pharmacotherapeutic Advisory Committee.

Determinations: The study variables will be evaluated at baseline and 3 months post-intervention. The primary variable is number of inappropriate prescriptions.

Statistical analysis: Percentage change will be measured before and after the intervention. Descriptive statistics will be performed for quantitative variables such as qualitative and comparison of means and proportions.

Expected results: Achieve a 10% decrease in inappropriate prescriptions

Applicability and Relevance: This study will expand the collaboration between the Pharmacy and Primary Care physicians, promoting the continuum of care, strengthening the safety culture, and improving prescribing habits.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Pharmacological treatment with at least one drug and for a period of more than three months

Exclusion Criteria:

* Individuals who at the time of the pharmaceutical review were in hospital
* Patients nearing the end of life
* Patients whose participation was considered by the doctor responsible to be potentially detrimental
* Patients not covered by the public healthcare or pharmacy system were excluded.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 862 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Drug-related problems | Basal
  Total count
Drug-related problems | Three months
  Total count
Drug-related problems | Basal
  average prm per patient
Drug-related problems | Three months
  average prm per patient
Drug-related problems | Basal
  % patients with prm
Drug-related problems | Three months
  % patients with prm
Polymedication: | Basal
  Average number of drugs
Polymedication: | Three months
  Average number of drugs
Polymedication: | Basal
  number of polymedicated patients (> 10 drugs)
Polymedication: | Three months
  number of polymedicated patients (>10 drugs)

SECONDARY OUTCOMES:
Sociodemographic variables | Basal
  genre: female/male
Sociodemographic variables | Basal
  median age
Sociodemographic variables | Basal
  average months in the geriatric residence
Description and classification of the DRPs detected Description and classification of the DRPs detected | Basal
  number of prm classified as indication
Description and classification of the DRPs detected Description and classification of the DRPs detected | Basal
  number of prm classified as adequate
Description and classification of the DRPs detected Description and classification of the DRPs detected | Basal
  number of prm classified as effectiveness
Description and classification of the DRPs detected Description and classification of the DRPs detected | Basal
  number of prm classified as security
Description and classification of the DRPs detected Description and classification of the DRPs detected | Three months
  number of prm classified as indication
Description and classification of the DRPs detected Description and classification of the DRPs detected | Three months
  number of prm classified as adequate
Description and classification of the DRPs detected Description and classification of the DRPs detected | Three months
  number of prm classified as effectiveness
Description and classification of the DRPs detected Description and classification of the DRPs detected | Three months
  number of prm classified as security

CONTACTS AND LOCATIONS:
Locations (1):
- Cecilia Campabadal Prats, Tarragona, Spain

REFERENCES:
- [Derived] Campabadal-Prats C, Aragones E, Romeu M, Salom-Garrigues C, Bejarano F, Martin Lujan F, Canadell L. Effectiveness of a structured pharmaceutical review of pharmacotherapeutic plans to reduce drug-related problems in nursing homes: a study protocol of a pragmatic quasi-experimental trial. Front Pharmacol. 2025 Jul 11;16:1522650. doi: 10.3389/fphar.2025.1522650. eCollection 2025. PMID 40717969